CLINICAL TRIAL: NCT07273734
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Ursodeoxycholic Acid Plus Lactulose vs Lactulose Alone for the Prevention of Overt Hepatic Encephalopathy After TIPS Placement
Brief Title: UDCA to Prevent Post-TIPS Hepatic Encephalopathy
Acronym: THEUDCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Kunming Medical University (Other); Qianjiang Central Hospital of Chongqing (Unknown); The Third People's Hospital of Kunming City (Unknown)
Responsible Party: Principal Investigator, Xiaoze Wang, Xiaoze Wang, MD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THE001
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Hepatic Encephalopathy (HE); TIPS
Keywords: TIPS; UDCA; Hepatic Encephalopathy (HE); Ursodeoxycholic acid
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Ursodeoxycholic Acid; Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UDCA + Lactulose (Experimental): Ursodeoxycholic acid (UDCA) 13-15 mg/kg/day orally, in divided doses (BID), starting ≤72 hours before TIPS and continued for 3 months. Lactulose syrup (25 mL BID) is initiated after TIPS procedure, titrated to achieve 1-2 soft stools per day, with stepwise dose reduction if diarrhea occurs.
  Interventions: Drug: Ursodeoxycholic Acid (UDCA); Drug: Lactulose
- Lactulose Alone (Active Comparator): Lactulose syrup (25 mL BID) is initiated after TIPS procedure, titrated to achieve 1-2 soft stools per day, with dose reduction as needed if diarrhea develops.
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Ursodeoxycholic Acid (UDCA) — 13-15 mg/kg/day orally, in divided doses (BID), starting ≤72 hours before TIPS and continued for 3 months.
  Arms: UDCA + Lactulose
Drug: Lactulose — Syrup 25 mL BID, initiated after TIPS procedure, titrated to 1-2 soft stools/day, with dose reduction if diarrhea occurs.

SUMMARY:
Hepatic encephalopathy (HE) commonly occurs after transjugular intrahepatic portosystemic shunt (TIPS). Ursodeoxycholic acid (UDCA) has been reported to alleviate neurodegenerative disease recently. This open-label multicenter randomized controlled trial tests whether adding UDCA (13-15 mg/kg/day) to standard lactulose prophylaxis reduces the incidence of overt HE (OHE; West Haven grade II-IV) after TIPS, compared with lactulose alone. The regimen starts within 72 hours before TIPS and continues for 3 months. The trial aims to evaluate the effect of UDCA in reducing the incidence of post-TIPS OHE.

DETAILED DESCRIPTION:
Post-TIPS OHE occurs in 35-50% of patients and worsens quality of life and resource use. Existing guidance consistently recommends lactulose as the backbone therapy for HE and for secondary prophylaxis, titrated to 2-3 soft stools/day; however, evidence for primary prophylaxis after TIPS has been limited and heterogeneous, and consensus varies across documents. Hydrophilic bile acids, especially ursodeoxycholic acid (UDCA), have demonstrated important anti-apoptotic and neuroprotective activities in clinical practice. Published experimental and clinical evidence suggests its potential therapeutic use as a disease-modifier in neurodegenerative and metabolic brain diseases. This trial evaluates whether bile-acid modulation with UDCA at standard hepatology dosing (13-15 mg/kg/day) combined with lactulose reduces early post-TIPS OHE. The protocol uses stratified randomization, prespecified outcome adjudication (West Haven), and intention-to-treat analysis. Key secondary endpoints include mortality, transplant-free survival, minimal HE tests (PHES, Stroop test), frailty, quality of life, and bile-acid/metabolomic profiling in optional sub-studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Confirmed cirrhosis (biopsy, elastography, or standard radiologic/biochemical criteria).
* Elective TIPS for (a) refractory/recurrent ascites and/or (b) recurrent variceal bleeding not responsive to treatment with endoscopic band ligation and beta-blockers.
* Preemptive TIPS for patients with variceal bleeding and Child-Pugh C (10-13 points), patients with Child-Pugh B and active bleeding during endoscopy, or patients with hepatic venous pressure gradient (HVPG) ≥ 20 mmHg.
* Ability to start study drug within 72 hours before TIPS.
* Signed informed consent.

Exclusion Criteria:

* Contraindications to TIPS (e.g., severe heart failure ≥NYHA III, severe pulmonary hypertension, uncontrolled sepsis, advanced HCC at risk with TIPS, unrelieved biliary obstruction, Child-Pugh score >13, main-trunk PVT if not recanalizable, technical infeasibility).
* Prior OHE grade II-IV without precipitating factor; overt neurological disease affecting cognition (e.g., Parkinson's, Alzheimer's).
* Current or planned ursodeoxycholic acid (UDCA) therapy for an approved indication (e.g., primary biliary cholangitis), or UDCA use within the prior 3 months.
* Current/recent rifaximin use (<3 months) or strong UDCA contraindication/hypersensitivity.
* Salvage TIPS.
* Non-cirrhotic portal hypertension.
* Pregnancy/lactation.
* Any condition that, in investigators' judgment, precludes safe participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Overt Hepatic Encephalopathy (OHE) within 3 Months After TIPS | From TIPS procedure (Day 0) to 3 months post-TIPS (Day 90).
  OHE defined as first occurrence of West Haven grade II-IV hepatic encephalopathy within 3 months after covered TIPS, adjudicated by investigator assessment according to West Haven criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maharshi S, Sharma BC. Prophylaxis of hepatic encephalopathy: current and future drug targets. Hepatol Int. 2024 Aug;18(4):1096-1109. doi: 10.1007/s12072-024-10647-9. Epub 2024 Mar 16. PMID 38492132
- [Result] Kronsten VT, Paintsil EK, Rodrigues S, Seager MJ, Bernal W, Shawcross DL. Hepatic Encephalopathy: When Lactulose and Rifaximin Are Not Working. Gastroenterology. 2025 Jun;168(6):1076-1084.e1. doi: 10.1053/j.gastro.2025.01.010. Epub 2025 Jan 24. No abstract available. PMID 39864468
- [Result] Djernes L, Vilstrup H, Ott P, Eriksen PL. Blood ammonia concentration measurement - effects of sampling site and cirrhosis during induced hyperammonaemia. Metab Brain Dis. 2024 Nov 20;40(1):21. doi: 10.1007/s11011-024-01442-4. PMID 39565434
- [Result] Shawcross DL, Thabut D, Amodio P. Ammonia - an enduring foe - What evaluating whole body ammonia metabolism can teach us about cirrhosis and therapies treating hepatic encephalopathy. J Hepatol. 2023 Aug;79(2):266-268. doi: 10.1016/j.jhep.2023.04.039. Epub 2023 May 12. No abstract available. PMID 37178732
- [Result] Wang X, Luo X, Yang L. Achieving an effective pressure reduction after TIPS: The need for a new target. J Hepatol. 2021 Jul;75(1):246-248. doi: 10.1016/j.jhep.2021.02.010. Epub 2021 Feb 20. No abstract available. PMID 33621635
- [Result] Wang X, Liu G, Wu J, Xiao X, Yan Y, Guo Y, Yang J, Li X, He Y, Yang L, Luo X. Small-Diameter Transjugular Intrahepatic Portosystemic Shunt versus Endoscopic Variceal Ligation Plus Propranolol for Variceal Rebleeding in Advanced Cirrhosis. Radiology. 2023 Aug;308(2):e223201. doi: 10.1148/radiol.223201. PMID 37606572
- [Result] Xiang Y, Tie J, Wang G, Zhuge Y, Wu H, Zhu X, Xue H, Liu S, Yang L, Xu J, Zhang F, Zhang M, Wei B, Li P, Wang Z, Wu W, Chen C, Yang S, Han Y, Tang C, Qi X, Zhang C. Post-TIPS Overt Hepatic Encephalopathy Increases Long-Term but Not Short-Term Mortality in Cirrhotic Patients With Variceal Bleeding: A Large-Scale, Multicenter Real-World Study. Aliment Pharmacol Ther. 2025 Apr;61(7):1183-1196. doi: 10.1111/apt.18509. Epub 2025 Feb 17. PMID 39962750
- [Result] Liu J, Ma J, Yang C, Chen M, Shi Q, Zhou C, Huang S, Chen Y, Wang Y, Li T, Xiong B. Sarcopenia in Patients with Cirrhosis after Transjugular Intrahepatic Portosystemic Shunt Placement. Radiology. 2022 Jun;303(3):711-719. doi: 10.1148/radiol.211172. Epub 2022 Mar 15. PMID 35289658
- [Result] Lv Y, Wang Q, Luo B, Bai W, Li M, Li K, Wang Z, Xia D, Guo W, Li X, Yuan J, Zhang N, Wang X, Xie H, Pan Y, Nie Y, Yin Z, Fan D, Han G. Identifying the optimal measurement timing and hemodynamic targets of portal pressure gradient after TIPS in patients with cirrhosis and variceal bleeding. J Hepatol. 2025 Feb;82(2):245-257. doi: 10.1016/j.jhep.2024.08.007. Epub 2024 Aug 22. PMID 39181214
- [Result] Ehrenbauer AF, Egge JFM, Gabriel MM, Tiede A, Dirks M, Witt J, Wedemeyer H, Maasoumy B, Weissenborn K. Comparison of 6 tests for diagnosing minimal hepatic encephalopathy and predicting clinical outcome: A prospective, observational study. Hepatology. 2024 Aug 1;80(2):389-402. doi: 10.1097/HEP.0000000000000770. Epub 2024 Feb 13. PMID 38349709
- [Result] Casadaban LC, Parvinian A, Minocha J, Lakhoo J, Grant CW, Ray CE Jr, Knuttinen MG, Bui JT, Gaba RC. Clearing the Confusion over Hepatic Encephalopathy After TIPS Creation: Incidence, Prognostic Factors, and Clinical Outcomes. Dig Dis Sci. 2015 Apr;60(4):1059-66. doi: 10.1007/s10620-014-3391-0. Epub 2014 Oct 15. PMID 25316553